CLINICAL TRIAL: NCT05616637
Title: Investigation of Inter-rater and Test-retest Reliability of Y Balance Test in Assessment of Dynamic Balance in Individuals With Pes Planus
Brief Title: Investigation of Inter-rater and Test-retest Reliability of Y Balance Test in Individuals With Pes Planus
Status: Completed | Type: Observational
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Istanbul Bilgi University (Other); Beykoz University (Other)
Responsible Party: Principal Investigator, Engin Caglar, Principal Investigator, Istanbul Gelisim University
Other Study IDs: PP002
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Flatfoot
Keywords: Postural Balance; Reproducibility of Results
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pes Planus: Participants with unilateral pes planus aged 18-40 years will be included in the study.
  Interventions: Diagnostic Test: Navicular Drop Test; Other: Lower Extremity Length Measurement; Other: Y Balance Test

INTERVENTIONS:
Diagnostic Test: Navicular Drop Test — While participants in sitting position, the navicular tuberosity (NT) will be palpated.The most distal protruding portion of the medial NT will be marked. Participants will be asked to stand with equal weight on both feet. The new distance will be measured. The navicular drop test (NDT) results will then be obtained by comparing the measured values between the sitting and standing positions. Each measurement will be repeated three times and the average of the 3 measurements will be calculated. The expression in mm of the distance between the two marks will be considered the amount of ND. The amount of navicular fall of 10 mm or more will be interpreted as pes planus. Measurements will be made on both extremities. As a result of the measurements, if pes planus is present in a single extremity, that extremity, if it is present in both extremities, the extremity with higher NDT or if it is equal on both sides, the dominant extremity will be tested.
Other: Lower Extremity Length Measurement — Lower extremity length will be recorded to normalize dynamic balance test data. The person will lie in the supine position. The distance between the umbilicus and the anterior superior of the spina iliaca will be measured in cm with the help of a tape measure. If there is no asymmetry, it will be assumed that there is no rotation in the pelvis, and it will be started to measure the length of the lower extremity. If pelvic asymmetry is detected, the pelvic position will be corrected manually. Then, the most inferior point of the spina iliaca anterior superior and the most distal point of the medial malleolus will be marked and measured and recorded. Lower extremity length and data in 3 different directions will be used in cm. The purpose of using formulas is to easily provide comparisons with other studies using the same type of data. The data obtained from the formula is expressed as a percentage of the length of the limb.
Other: Y Balance Test — While the individual tries to balance on one bare foot at the midpoint of the assembly, the individual will also be asked to reach as far as possible with the other foot in the anterior, posteromedial and posterolateral directions, touch the tip of the toe, and then immediately return to the starting position without disturbing the balance. The test will be evaluated for 3 repetitions. Situations where the participant will be requested to repeat the test: the foot on the ground passes the reference point or the heel lifts off the ground, perturbations caused by the environment, contact of the foot with the ground, and loss of balance when returning to the starting position. 10 seconds between 3 repetitions during testing will be given. Each participant will be given the right to try 6 times before starting the test in order to eliminate the possible learning parameter. The test will be repeated 3 times in each direction and the closest distance in cm will be recorded.

SUMMARY:
Pes Planus is characterized by the descent of the medial longitudinal arch, eversion of the hindfoot, and dorsiflexion and abduction of the midfoot. Disorders in the bones of the foot, dysfunction of the tibialis posterior muscle, shortness of the Achilles tendon or weakness in the muscles may pose a risk for pes planus.

In a study in which 80 female participants aged 65 and over participated voluntarily, it was shown that 90% of the deformities seen in the foot were pes planus. In another study conducted with adults aged 18-21 years, pes planus was found with a rate of 13.6%. In a study in a group of 500 people aged 18-25 years, this rate was found to be 29%.

Since exercise, physical activity and walking for a long time will cause foot and leg pain in people with pes planus, the level of physical activity of these people may be limited. There are studies examining the relationship between pes planus and different physical parameters. It has been determined as a result of some studies that the balance, which is one of these parameters, is negatively affected by the presence of pes planus.

According to the literature, many studies have used the Y test in the evaluation of dynamic balance in individuals with pes planus. However the reliability of the Y Balance Test, which is a valid and reliable method for assessing balance in healthy individuals, has not been found in individuals with pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being between the ages of 18-40,
* Having pes planus.

Exclusion Criteria:

* Having had lower extremity or spine surgery,
* Having a neurological or rheumatic disease,
* Having a problem with vision and hearing,
* Having suffered a lower extremity injury in the last 1 year,
* Presence of acute or chronic pain,
* Regular participation in sports activities,
* Being pregnant,
* Ambulation with an assistive device,
* Active participation in treatment,
* Presence of lower extremity inequality.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Young adults aged 18-40, with pes planus and volunteering to participate in the study will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Y Balance Test | Baseline
  Dynamic Balance Test

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JA, Lim OB, Yi CH. Difference in static and dynamic stability between flexible flatfeet and neutral feet. Gait Posture. 2015 Feb;41(2):546-50. doi: 10.1016/j.gaitpost.2014.12.012. Epub 2014 Dec 22. PMID 25560044
- [Background] Kim EK, Kim JS. The effects of short foot exercises and arch support insoles on improvement in the medial longitudinal arch and dynamic balance of flexible flatfoot patients. J Phys Ther Sci. 2016 Nov;28(11):3136-3139. doi: 10.1589/jpts.28.3136. Epub 2016 Nov 29. PMID 27942135
- [Background] Alam F, Raza S, Moiz JA, Bhati P, Anwer S, Alghadir A. Effects of selective strengthening of tibialis posterior and stretching of iliopsoas on navicular drop, dynamic balance, and lower limb muscle activity in pronated feet: A randomized clinical trial. Phys Sportsmed. 2019 Sep;47(3):301-311. doi: 10.1080/00913847.2018.1553466. Epub 2018 Dec 5. PMID 30517043
- [Background] Alshehre Y, Alkhathami K, Brizzolara K, Weber M, Wang-Price S. Reliability and Validity of the Y-balance Test in Young Adults with Chronic Low Back Pain. Int J Sports Phys Ther. 2021 Jun 1;16(3):628-635. doi: 10.26603/001c.23430. PMID 34123515